CLINICAL TRIAL: NCT06895759
Title: AVA-CO2-R: Impact of CO2 Absorption on Gas Exchange and Ventilation Patterns While Breathing Into a Snow Air Pocket - An Experimental Study
Brief Title: Impact of CO2 Absorption on Gas Exchange and Ventilation Patterns While Breathing Into a Snow Air Pocket
Acronym: AVACO2R
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Eurac
Record Dates: First submitted 2025-03-14; First posted 2025-03-26 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Avalanche Burial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breathing with soda lime (Experimental): Respiration into a snow air pocket through an experimental rebreathing circuit with the integration of a soda lime canister.
  Interventions: Device: Soda lime
- Breathing without soda lime (Sham Comparator): Respiration into a snow air pocket through an experimental rebreathing circuit without the integration of a soda lime canister.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Soda lime — Respiration into a snow air pocket through an experimental rebreathing circuit with the integration of a soda lime canister.
  Arms: Breathing with soda lime
Device: Sham — Respiration into a snow air pocket through an experimental rebreathing circuit without the integration of a soda lime canister.
  Arms: Breathing without soda lime

SUMMARY:
Asphyxia is by far the most common cause of death after critical avalanche burial. The presence of an air pocket increases the survival chances, but expired air rich in carbon dioxide (CO2) progressively displaces oxygen (O2) in the air pocket, a phenomenon known as displacement asphyxia. In addition, an increase in the inspired concentration of CO2 (FiCO2) reduces the alveolar partial pressure of O2 (PAO2), as explained by the alveolar gas equation. Underlining this, a recent experimental porcine study showed that an increased FiCO2 is the leading cause of the decrease in PaO2. By removing CO2 in an experimental avalanche burial, normoxia persisted even after 90 minutes of burial, while, in the absence of CO2 removal, hypoxemia and hypercapnia occurred after only 10 minutes. Additionally, hypercapnia increases pulmonary vascular resistance, reduces cardiac output and can lead to life-threatening hemodynamic instability. Hypercapnia can speed up the cooling rate, and the combination of hypothermia with hypoxia and hypercapnia may result in a worse neurological outcome in completely buried avalanche patients compared to patients suffering solely hypothermic cardiac arrest.

Taken together, these findings suggest that removing CO2 from the air-pocket could prevent, or at least delay, the hypercapnic condition with its deleterious consequences and consequently increase the survival after complete avalanche burial.

The main aim of the study is to investigate the effectiveness of soda lime in removing CO2 while breathing into a snow air pocket, and to assess its impact on gas exchange, ventilation patterns, and hemodynamics.

DETAILED DESCRIPTION:
Introduction

Background and aims

Asphyxia is by far the most common cause of death after critical avalanche burial. The presence of an air pocket increases the survival chances , but expired air rich in carbon dioxide (CO2) progressively displaces oxygen (O2) in the air pocket, a phenomenon known as displacement asphyxia. In addition, an increase in the inspired concentration of CO2 (FiCO2) reduces the alveolar partial pressure of O2 (PAO2), as explained by the alveolar gas equation. Underlining this, a recent experimental porcine study showed that an increased FiCO2 is the leading cause of the decrease in PaO2. By removing CO2 in an experimental avalanche burial, normoxia persisted even after 90 minutes of burial, while, in the absence of CO2 removal, hypoxemia and hypercapnia occurred after only 10 minutes. Additionally, hypercapnia increases pulmonary vascular resistance, reduces cardiac output and can lead to life-threatening hemodynamic instability. Hypercapnia can speed up the cooling rate, and the combination of hypothermia with hypoxia and hypercapnia may result in a worse neurological outcome in completely buried avalanche patients compared to patients suffering solely hypothermic cardiac arrest.

Taken together, these findings suggest that removing CO2 from the air-pocket could prevent, or at least delay, the hypercapnic condition with its deleterious consequences and consequently increase the survival after complete avalanche burial.

The main aim of the study is to investigate the effectiveness of soda lime in removing CO2 while breathing into a snow air pocket, and to assess its impact on gas exchange, ventilation patterns, and hemodynamics.

Study endpoints

Primary endpoints:

* Time to reach an end-tidal CO2 (etCO2) of 70 mmHg or partial pressures of carbon dioxide in arterial blood (PaCO2) of 65 mmHg
* Difference in etCO2 and PaCO2 either after 60 minutes (i.e. maximum test duration) or at test interruption

Secondary endpoints:

* Time to reach an oxygen saturation (SpO2) ≤75%
* Time to reach partial pressures of oxygen in arterial blood (PaO2) ≤ 45 mmHg
* Differences in O2 consumption (VO2), CO2 production (VCO2)
* Differences in inspiratory fraction of CO2 (FiCO2) and O2 (FiO2)
* Differences in concentrations CO2 and O2 in the air pocket
* Difference in ventilatory patterns [minute ventilation (VE), tidal volume (TV), respiratory rate (RR), work of breathing]
* Difference in blood pressure (BP), cardiac output (CO) and heart rate (HR)
* Difference in left and right ventricular strain measured by echocardiography
* Difference in cerebral blood flow

Methods

Study design Interventional, non-pharmacological study on healthy volunteers with a randomized, cross-over design.

Participants will breathe into a 0.5-liter snow air pocket using an experimental rebreathing circuit. Each participant will complete the test twice-once with soda lime integrated into the circuit and once without (crossover design). The order of the tests will be randomized, with a 60-minutes wash-out period between them.

Subject number: about 20 participants will be included.

Inclusion criteria

* Age: 18 - 60 yrs
* Body mass index < 30 kg/m2
* ASA class ≤2
* providing informed and written consent Exclusion criteria
* ASA class >2
* Pregnancy
* Smoking

Protocol After having received a detailed explanation of the study's purpose and procedures, participants will be required to provide informed written consent. Subsequently, a physician from the study team will conduct a general medical examination.

Participants will breathe into a 0,5-liter snow air pocket using an experimental rebreathing circuit. Each participant will complete the test twice-once with soda lime integrated into the circuit and once without (crossover design). The order of the tests will be randomized, with a wash-out period of 60 minutes between them.

The rebreathing circuit will be connected to a snow air-pocket with a total capacity of 0,5 liters. A two-way non-rebreathing valve and several sensors will be integrated into the breathing circuit in order to allow the measurement of respiratory rate (RR), tidal volume (VT) and minute ventilation (VE), oxygen consumption (VO2), carbon dioxide production (VCO2), inspiratory and expiratory respiratory gas concentrations [i.e. fractional content of inspired oxygen (FiO2), fractional content of inspired carbon dioxide (FiCO2), fractional content of expired oxygen (FeO2), fractional content of expired carbon dioxide (FeCO2)]. A capnograph will be located in the expiratory part of the breathing circuit to allow the measurement of the end-tidal carbon dioxide (etCO2) over time. O2 and CO2 concentration in the air pocket will also be measured. Participants will then be instrumented with an arterial catheter, placed in the radial artery, to record arterial blood pressure and cardiac output continuously and to allow for arterial blood drawings. An esophageal balloon catheter placed transnasally in the lower two thirds of the intrathoracic esophagus and connected to a dedicated monitoring device will allow to measure the esophageal pressure swings and to calculate the of work of breathing. In addition, an electrocardiogram and a pulse oximeter will be placed to monitor the vital parameters of the subjects over time. Left and right ventricular strain will be measured with echocardiography and cerebral blood flow will be quantified by transcranial doppler ultrasound.

Subsequently, the subject will be placed in left lateral position and baseline measurements will be taken, including respiratory rate (RR), tidal volume (TV), minute ventilation (MV), etCO2, paO2 and paCO2, VO2, VCO2, esophageal pressure swings, blood pressure (BP), cardiac output (CO), heart rate (HR), transcranial doppler and echocardiographic parameters.

The test will run for a maximum of 35 minutes. It will be terminated earlier if any of the following interruption criteria are met:

* Duration of 35 min reached
* SpO2 ≤75%
* etCO2 ≥ 70 mmHg or PaCO2 ≥65 mmHg
* Participant request to interrupt the study

During the test, the following parameters will be measured continuously: RR, TV, MV, etCO2, paO2 and paCO2, VO2, VCO2, esophageal pressure swings, BP, HR and CO. Additionally, transcranial Doppler ultrasound and echocardiography will be performed at regular intervals, along with arterial blood gas analysis. Measures will be continued for few minutes after test termination.

After a 60-minutes wash-out period, participants will undergo the second test (crossover design).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 60 yrs.
* Body mass index < 30 kg/m2
* ASA class ≤2
* Providing informed and written consent

Exclusion Criteria:

* ASA >2
* Pregnancy
* Smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to reach an end-tidal CO2 or partial pressures of carbon dioxide in arterial blood (PaCO2) | 35 minutes
  Time to reach an end-tidal CO2 (etCO2) of 70 mmHg or partial pressures of carbon dioxide in arterial blood (PaCO2) of 65 mmHg
Time to reach an oxygen saturation (SpO2) | 35 minutes
  Time to reach an oxygen saturation (SpO2) ≤75%

SECONDARY OUTCOMES:
Difference in end-tidal CO2 (etCO2) and partial pressures of carbon dioxide in arterial blood (PaCO2) | 35 minutes
  Difference in end-tidal CO2 (etCO2) and partial pressures of carbon dioxide in arterial blood (PaCO2) between the intervention and control during the test
Partial pressure of oxygen | 35 minutes
  Time to reach partial pressures of oxygen in arterial blood (PaO2) ≤ 45 mmHg
Differences in inspiratory fraction of CO2 (FiCO2) and O2 (FiO2) | 35 minutes
  Differences in inspiratory fraction of CO2 (FiCO2) and O2 (FiO2) between the intervention and control during the test
Difference in minute ventilation (VE) | 35 minutes
  Difference in minute ventilation (VE) during the test between the intervention and control
Difference in cardiac output (CO) | 35 minutes
  Difference in cardiac output (CO) between the intervention and control during the test
Difference in left and right ventricular strain | 35 minutes
  Difference in left and right ventricular strain measured by echocardiography between the intervention and control during the test
Difference in cerebral blood flow | 35 minutes
  Difference in cerebral blood flow between the intervention and control during the test
Difference in cerebral oxygen saturation | 35 minutes
  Difference in cerebral oxygen saturationbetween the intervention and control during the test
Difference in work of breathing | 35 minutes
  Difference in work of breathing (WOB) during the test between the intervention and control. WOB is calculated by integrating tidal volume with esophageal pressure (measured via an esophageal balloon) during inspiration, and is expressed in Joules.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rauch, MD, PhD, Principal Investigator — Eurac research, Institute of Mountain Emergency Medicine
Locations (1):
- terraXCube, Bolzano, Italy/BZ, Italy

IPD SHARING:
Plan to Share IPD: No